CLINICAL TRIAL: NCT04785937
Title: Accuracy of Imaging Techniques Including Ultrasound and Magnetic Resonance Imaging in the Diagnosis of Steatohepatitis and Fibrosis in Patients With Non-Alcoholic Fatty Liver Disease: Comparison With the Histological Reference Standard
Brief Title: Accuracy of Imaging Techniques in Diagnosing Steatohepatitis and Fibrosis in NAFLD Patients
Acronym: ImagingNAFLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 859/2018/SPER/AUSLRE
Record Dates: First submitted 2021-02-28; First posted 2021-03-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Steatohepatitis, Nonalcoholic; Liver Fibroses
Keywords: Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Diagnostic Ultrasound; Biopsy; Non-Inferiority Trial
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Ultrasonography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging and Biopsy (Experimental): All patients undergo both liver biopsy and liver imaging (US and MR) to assess the diagnostic performance of imaging compared to histopathological examination in the diagnosis of NASH and fibrosis.
  Interventions: Diagnostic Test: Ultrasound and Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Ultrasound and Magnetic Resonance — liver ultrasound (US), including shear wave elastography (SWE) with liver stiffness measurement and US- fatty liver indicator (US-FLI), and a multiparametric unenhanced liver magnetic resonance examination including MR spectroscopy (MRS), Proton Density Fat Fraction (PDFF) and T2* measurement with Multiecho technique, T1 mapping with Inversion Recovery method, and Intravoxel Incoherent Motion diffusion weighted imaging (IVIM-DWI), measuring different parameters.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a highly prevalent condition, and when fatty liver is associated with inflammation and hepatocellular injury (steatohepatitis), it can lead to fibrosis, cirrhosis, liver failure and hepatocellular carcinoma. Liver biopsy is the gold standard for NAFLD assessment but has several drawbacks. Several drugs for NASH are now in phase 2-3 trials, and if medical treatments become available, non-invasive tools to identify patients who may benefit from a therapeutic intervention will be strongly needed. Some imaging methods have shown promising potential in fibrosis and NASH diagnosis. This study aims to evaluate the diagnostic accuracy of non-invasive imaging methods, including ultrasound (US) and Magnetic Resonance (MR) techniques, in diagnosing NASH and fibrosis in patients with or at high risk of NAFLD, using liver biopsy as the reference standard. Consecutive patients with a clinical indication for liver biopsy assessment of NAFLD are enrolled in this non-inferiority study. They undergo both a liver US and a multiparametric unenhanced liver MR examination. As reference standard, histological diagnosis of fibrosis and steatohepatitis made according to the fatty liver inhibition of progression (FLIP) algorithm is used. Sensitivity and specificity of imaging parameters alone or in different combinations will be calculated with the aim of finding one or more tests with at least 90% sensitivity/specificity compared to liver biopsy.

DETAILED DESCRIPTION:
The estimated overall global prevalence of non-alcoholic fatty liver disease (NAFLD) is around 25% and projected at 33.5% in 2030. While simple steatosis without evidence of inflammation and hepatocellular injury (non-alcoholic fatty liver) is generally a benign condition, non-alcoholic steatohepatitis (NASH) can progress to fibrosis, cirrhosis, liver failure and hepatocellular carcinoma. Since only histological analysis can accurately evaluate NAFLD patterns, liver biopsy is the gold standard for assessment, and it should be considered in patients who are at increased risk of having steatohepatitis and/or fibrosis. Major drawbacks are its invasive nature, risk of complications, sampling errors and inter and intra-observer variability. Currently, there are no approved therapies for NASH. However, several drugs are now in phase 2 and 3 trials, and results are expected in 1-2 years. If medical treatments become available, screening for steatohepatitis and fibrosis will be recommended in high-risk patients. The lack of non-invasive tools to identify patients who may benefit from a therapeutic intervention is a central issue. Should liver biopsy be avoided or reserved for a more limited number of undetermined or high-risk patients, the benefit-harm balance of NASH screening and therapies would undergo a major change. Some imaging methods, mostly ultrasound (US) or Magnetic Resonance (MR) techniques, have shown promising potential in fibrosis and NASH diagnosis.

The objective of this study is to evaluate the diagnostic accuracy of non-invasive imaging techniques including US and MR methods, in diagnosing NASH and fibrosis in patients with or at high risk of NAFLD, using liver biopsy as the reference standard.

Consecutive patients with a clinical indication for liver biopsy assessment of NAFLD are enrolled in this non-inferiority study. They undergo both a liver ultrasound (US), including shear wave elastography (SWE) with liver stiffness measurement and US- fatty liver index (US-FLI), and a multiparametric unenhanced liver magnetic resonance examination including MR spectroscopy (MRS), Proton Density Fat Fraction (PDFF) and T2* measurement with Multiecho technique, T1 mapping with Inversion Recovery method, and Intravoxel Incoherent Motion diffusion weighted imaging (IVIM-DWI), measuring different parameters. As reference standard, histological diagnosis of fibrosis and steatohepatitis made according to the fatty liver inhibition of progression (FLIP) algorithm is used. Sensitivity and specificity of imaging parameters alone or in different combinations will be calculated, with the aim of finding one or more tests with at least 90% sensitivity/specificity compared to liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* clinical indication to perform a liver biospy for NAFLD assessment based on all of the following:

  1. presence of liver steatosi at ultrasound
  2. at least one risk factor for NASH/fibrosis (obesity, or type 2 diabetes mellitus, or metabolic syndrome)
  3. increased liver enzymes (at least one of: GOT>40 U/l, GPT>49 U/l, GGT>75 U/l) or high NAFLD fibrosis score (>0.675), or intermediate NAFLD fibrosis score (between -1.455 and 0.675) and increased liver stiffness at transient elastography (>7 KPa).
* consent to participate in the study

Exclusion Criteria:

* age < 18 years
* secondary causes of liver steatosis (moderate to severe alcohol consumption, steatogenic drugs)
* known diffuse liver diseases other than NAFLD (cirrhosis, viral or autoimmune hepatitis, hemochromatosis, amiloidosis, other) or previous primary or secondary liver neoplasms
* contraindications to perform liver biopsy (ascites, platelet count<50.000/mmc, INR>1.5, PT>50%, serum bilirubin >3 mg/dL)
* contraindications to perform magnetic resonance (pace-maker, claustrophobia, pregnancy, MR-unsafe metallic implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
False positives | baseline
  false positives of each imaging parameter compared to liver biopsy in the diagnosis of NASH/fibrosis
False negatives | baseline
  false negatives of each imaging parameter compared to liver biopsy in the diagnosis of NASH/fibrosis
Sensitivity | baseline
  Sensitivity of each imaging parameter compared to liver biopsy in the diagnosis of NASH/fibrosis
Specificity | baseline
  Specificity of each imaging parameter compared to liver biopsy in the diagnosis of NASH/fibrosis

SECONDARY OUTCOMES:
Correlation of quantitative imaging parameters with histopathological, demographic, anthropometric and clinical characteristics | baseline
  Correlation of imaging parameters (US-FLI, US-SWE, MR-PDFF, MR-T1, MR-T2*, MR-IVIM coefficients, MRS metabolites) with histopathological (percentage of steatosis, lobular inflammation, hepatocellular ballooning, fibrosis), demographic (age, sex), anthropometric (BMI, waist circumference) and clinical (liver enzymes, NAFLD fibrosis score, FIB4) characteristics
Number of patients whit incomplete or unreliable imaging tests | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Pattacini, MD, Study Director — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Sumida Y, Nakajima A, Itoh Y. Limitations of liver biopsy and non-invasive diagnostic tests for the diagnosis of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. World J Gastroenterol. 2014 Jan 14;20(2):475-85. doi: 10.3748/wjg.v20.i2.475. PMID 24574716
- [Background] Issa D, Patel V, Sanyal AJ. Future therapy for non-alcoholic fatty liver disease. Liver Int. 2018 Feb;38 Suppl 1:56-63. doi: 10.1111/liv.13676. PMID 29427492
- [Background] Park CC, Nguyen P, Hernandez C, Bettencourt R, Ramirez K, Fortney L, Hooker J, Sy E, Savides MT, Alquiraish MH, Valasek MA, Rizo E, Richards L, Brenner D, Sirlin CB, Loomba R. Magnetic Resonance Elastography vs Transient Elastography in Detection of Fibrosis and Noninvasive Measurement of Steatosis in Patients With Biopsy-Proven Nonalcoholic Fatty Liver Disease. Gastroenterology. 2017 Feb;152(3):598-607.e2. doi: 10.1053/j.gastro.2016.10.026. Epub 2016 Oct 27. PMID 27911262
- [Background] Besutti G, Valenti L, Ligabue G, Bassi MC, Pattacini P, Guaraldi G, Giorgi Rossi P. Accuracy of imaging methods for steatohepatitis diagnosis in non-alcoholic fatty liver disease patients: A systematic review. Liver Int. 2019 Aug;39(8):1521-1534. doi: 10.1111/liv.14118. Epub 2019 May 8. PMID 30972903
- [Background] Ballestri S, Lonardo A, Romagnoli D, Carulli L, Losi L, Day CP, Loria P. Ultrasonographic fatty liver indicator, a novel score which rules out NASH and is correlated with metabolic parameters in NAFLD. Liver Int. 2012 Sep;32(8):1242-52. doi: 10.1111/j.1478-3231.2012.02804.x. Epub 2012 Apr 22. PMID 22520641
- [Background] Eddowes PJ, McDonald N, Davies N, Semple SIK, Kendall TJ, Hodson J, Newsome PN, Flintham RB, Wesolowski R, Blake L, Duarte RV, Kelly CJ, Herlihy AH, Kelly MD, Olliff SP, Hubscher SG, Fallowfield JA, Hirschfield GM. Utility and cost evaluation of multiparametric magnetic resonance imaging for the assessment of non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2018 Mar;47(5):631-644. doi: 10.1111/apt.14469. Epub 2017 Dec 22. PMID 29271504
- [Background] Pavlides M, Banerjee R, Tunnicliffe EM, Kelly C, Collier J, Wang LM, Fleming KA, Cobbold JF, Robson MD, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging for the assessment of non-alcoholic fatty liver disease severity. Liver Int. 2017 Jul;37(7):1065-1073. doi: 10.1111/liv.13284. Epub 2017 May 30. PMID 27778429
- [Background] Bedossa P; FLIP Pathology Consortium. Utility and appropriateness of the fatty liver inhibition of progression (FLIP) algorithm and steatosis, activity, and fibrosis (SAF) score in the evaluation of biopsies of nonalcoholic fatty liver disease. Hepatology. 2014 Aug;60(2):565-75. doi: 10.1002/hep.27173. Epub 2014 Jun 26. PMID 24753132